CLINICAL TRIAL: NCT05844969
Title: Circle Method Observational Project - Non-interventional, Retrospective, Multicenter Data Collection to Validate Circle Method for Sizing and Positioning in Bicuspid Aortic Valves
Brief Title: Circle Method Observational Project - Non-interventional, Retrospective, Multicenter Data Collection
Status: Not yet recruiting | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: CMOP
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Aortic Stenosis With Bicuspid Valve

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this non-interventional, retrospective data analysis is to validate the circle method for patients with bicuspid aortic heart valves undergoing transcatheter aortic heart valve implantation (TAVI).

The main aims are:

* to assess whether patients with bicuspid aortic valves that received a TAVI suffered from fewer complications

  * if valve size was identical to the one determined using the circle method compared to
  * a case where circle method derived valve size is different from the actually implanted valve
* to develop recommendations on how to size the valve using the circle method.

DETAILED DESCRIPTION:
The bicuspid aortic valve (BAV) is the most common heart valve abnormality and is associated with a number of cardiac complications, including infective endocarditis, aortic dissection, aortic dilatation, and the development of severe aortic stenosis (AS). Due to its anatomical characteristics BAV has been considered a contraindication to transcatheter aortic valve implantation (TAVI), a standard treatment of AS. However, several recent trials have presented promising results indicating TAVI to be a safe alternative to surgery for low risk patients and more patients with BAV have been considered for TAVI.

There are several sizing techniques for TAVI in BAV, including an annular sizing, a supra-annular sizing, and a balloon sizing, yet there is still no consensus on the most appropriate technique. Although annular sizing remains the major approach in most patients with BAV, some BAV anatomies may profit from the supra-annular sizing. Recently published consensus for sizing and positioning the balloon-expandable Edwards SAPIEN 3 transcatheter heart valve (THV) in BAV describes the anatomical features that influence sizing optimization. The novel circle technique has also been proposed in the presence of the unique anatomical factors and sizing at the supra-annular level. This method is particularly helpful for visually identifying anatomic features, indicating the sealing zone at the commissures, visually reassuring of the size and position, and treating patients with large annuli. Currently, there are limited data validating the circle method for identifying sizing and positioning for TAVI in BAV patients.

In this non-interventional, retrospective, multicenter data collection and analysis we aim to validate the circle method for sizing and positioning in bicuspid aortic valves.

Due to the non-interventional character of the project, no additional burden will be put on the patients eligible for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bicuspid aortic valves who underwent aortic valve replacement with a balloon expandable valve (SAPIEN 3 / Ultra)
* Computed Tomography data available

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with bicuspid valve disease who underwent aortic valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Complications | 12 months
  To assess whether patients with bicuspid aortic valves that received a SAPIEN 3 / Ultra THV suffered from fewer complications
  * if valve size was identical to the one determined using the circle method compared to
  * a case where circle method derived valve size is different from the actually implanted valve

SECONDARY OUTCOMES:
Sizing with Circle Method | 12 months
  To develop recommendations on how to size the valve using the circle method.

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Costanzo, Dr., Study Director — Royal Papworth Hospital NHS Foundation Trust; Ioannis Lianos, Dr., Principal Investigator — Guy's and St Thomas NHS Foundation Trust; Tiffany Patterson, Dr., Principal Investigator — Guy's and St Thomas NHS Foundation Trust; Timothy Bagnall, Dr., Principal Investigator — University Hospitals Sussex NHS Foundaton Trust; Angie Ghattas, Dr., Principal Investigator — Golden Jubilee National Hospital
Locations (4):
- United Kingdom (4):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Golden Jubilee National Hospital, Clydebank
  - Guy's and St Thomas NHS Foundation Trust, London
  - University Hospitals Sussex NHS Foundation Trust, Worthing

IPD SHARING:
Plan to Share IPD: No
Only anonymized, aggregated data will be shared.